CLINICAL TRIAL: NCT03660293
Title: Prediction and Prevention of Asymptomatic Cardiovascular Insult in Type 1 Diabetic Children: Comparative Effectiveness of Cardio-protective Drugs
Brief Title: Prediction and Prevention of Asymptomatic Cardiovascular Insult in Type 1 Diabetic Children: Comparative Effectiveness of Cardioprotective Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rasha Mohamed Gamal, Ass. Professor of Pediatrics, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 31499/04/17
Record Dates: First submitted 2018-07-11; First posted 2018-09-06 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Atorvastatin; Captopril; Carnitine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- diabetic- no cardioprotectives (No Intervention): 25 child with type 1 diabetes mellitus will not receive any cardio protective drug
- diabetic-Atorvastatin (Experimental): 25 child with type 1 diabetes mellitus will receive Statin (2 mg/kg/day)
  Interventions: Drug: Atorvastatin
- diabetic-Captopril (Experimental): 25 child with type 1 diabetes mellitus will receive Captopril (0.2 mg/kg/day)
  Interventions: Drug: Captopril
- diabetic-L-Carnitine (Experimental): 25 child with type 1 diabetes mellitus will receive L-carnitine (50 mg/kg/day)
  Interventions: Drug: L-carnitine
- Controls (No Intervention): 50 healthy children, of matched age and sex, with no symptoms of cardiac diseases

INTERVENTIONS:
Drug: Atorvastatin — cardio-protective agents
  Arms: diabetic-Atorvastatin
Drug: Captopril — cardio-protective agents
  Arms: diabetic-Captopril
Drug: L-carnitine — cardio-protective agents
  Arms: diabetic-L-Carnitine

SUMMARY:
Diabetic cardiomyopathy (DCM) is a distinct clinical entity of diabetic heart muscle that describes diabetes associated changes in the structure and function of the myocardium in the absence of coronary artery disease, hypertension, and valvular disease. Oxidative stress plays a critical role in DCM development. DCM can be diagnosed using the novel methods of echocardiography (tissue Doppler imaging, Speckling tracking techniques and more recent real time 4D echocardiography). There is a possible cardioprotective effect of statins, Captopril and L-Carnitine in type 1 diabetic children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescent suffering from type 1 Diabetes Mellitus, for at least 3 years from the onset of the disease.

Exclusion Criteria:

* Children with Congenital Heart Diseases.
* Children with acquired cardiac diseases.
* Children with other systemic diseases.
* Symptomatic diabetic cardiomyopathy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The cardiac changes induced by Simvastatin, captopril and L-Carnitine in type 1 diabetic children and adolescents. | before and after 4 months of receiving cardio-protective agents
  Corrected QT interval(QTc) and QT dispersion in ElectroCardioGram
The cardiac changes induced by Simvastatin, captopril and L-Carnitine in type 1 diabetic children and adolescents. | before and after 4 months of receiving cardio-protective agents
  Left Ventricular End Systolic Volume (ml). Left Ventricular End Diastolic Volume (ml). Ejection Fraction (EF %) and left ventricular strain using echocardiography.

SECONDARY OUTCOMES:
The role of Troponin I levels as a cardiac marker for detection of asymptomatic cardiovascular insult in diabetic children. | first day
  Serum Cardiac troponin I by Enzyme Linked ImmunoSorbant Assay
The role of recent echocardiographic parameters for early detection of silent myocardial dysfunction | first day
  Echocardiography
Identification of risk factors for developing diabetic cardiac insult. | first day

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Derived] Badreldeen A, El Razaky O, Erfan A, El-Bendary A, El Amrousy D. Comparative study of the efficacy of captopril, simvastatin, and L-carnitine as cardioprotective drugs in children with type 1 diabetes mellitus: a randomised controlled trial. Cardiol Young. 2021 Aug;31(8):1315-1322. doi: 10.1017/S1047951121000226. Epub 2021 Feb 4. PMID 33536102